CLINICAL TRIAL: NCT06714682
Title: Ultrasound-Guided Modified Pectoral Plane (PECS II) Block Versus Erector Spinae Plane Block (ESPB) for Postoperative Analgesia of Modified Radical Mastectomy
Brief Title: Comparing Post-operative Analgesia After (PECS II) Block and (ESPB) in Modified Radical Mastectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, mohamed ibrahim hassan mohamed, lecturer of anesthesia, intensive care and pain management, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FMASU MS458/2024
Record Dates: First submitted 2024-11-28; First posted 2024-12-04 (Actual); Results first posted 2025-05-04 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Anaesthesia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ultrasound-Guided Modified Pectoral Plane Block group (Active Comparator): first group 10 patients
  Interventions: Procedure: Modified Pectoral Plane block group
- Erector Spinae Plane Block group (Active Comparator): second group 10 patients
  Interventions: Procedure: Erector spinae plane block group.

INTERVENTIONS:
Procedure: Modified Pectoral Plane block group — The patient will lay supine with the ipsilateral arm abducted and externally rotated and the elbow flexed at 90 degrees. The probe will be placed transversely between the clavicle medially and above and the shoulder joint laterally. After identifying the pectoralis major and minor muscles and the plane between them, the probe will be pushed 1-2 cm caudally and medially. In a caudal tilt, within a biconvex space, the artery will be recognised. After that, the block needle will be inserted in an in-plane approach to the artery's location and 10 mL of 0.25% bupivacaine will be administered Then probe will be moved laterally and caudally towards the anterior axillary fold until the serratus muscle appears beneath the pectoralis minor muscle attaching to the underlying ribs. The needle will target the plane between pectoralis minor and serratus muscles at the level of the third rib, followed by negative aspiration into the fascial plane then injection of 10 mL of 0.25 bupivacaine.
  Other Names: PECS II
  Arms: Ultrasound-Guided Modified Pectoral Plane Block group
Procedure: Erector spinae plane block group. — The block will be performed with the patient in a sitting position , The high-frequency linear probe will be placed in a longitudinal orientation 3 cm from the midline. Once the erector spinae muscle and the transverse processes identified, the block needle will be inserted in a caudad-to-cephalad direction until the tip lay in the interfacial plane deep to the erector spinae muscle, 20 mL of 0.25% bupivacaine will be administered for block performance.
  Other Names: ESPB
  Arms: Erector Spinae Plane Block group

SUMMARY:
The aim of this study is to compare the analgesic efficacies of the modified pectoral plane block (PECS II) and the erector spinae plane block (ESPB) after modified radical mastectomy surgery through assessment of post-operative pain severity by Visual Analogue Score at PACU as a primary outcome and at 2 hours, 4 hours, 8 hours, 12 hours, 18 hours and 24 hours post-operatively also by comparing time of first rescue analgesia and cumulative post-operative meperidine consumption in the first 24 hours as secondary outcomes.

DETAILED DESCRIPTION:
During MRM , some of the nerves in the chest are affected so most women have some level of pain in the days after the procedure. Severe acute postoperative pain following breast surgery is an independent risk factor in the development of chronic post-mastectomy pain , not only increasing the risk of persistent agony and prolongs hospitalization, it also affects recovery and increases healthcare costs .

Multimodal techniques for pain management have been recommended by the American Society of Anesthesiologists (ASA) for the management of acute postoperative pain . These techniques include oral analgesics as opioids, paracetamol and nonsteroidal anti inflammatory drugs (NSAIDs) , intravenous (IV) and regional analgesia. Inappropriate postoperative analgesia may increase morbidity and mortality .

PECS-II block is an interfascial plane block in which local anesthetic is injected between serratus anterior and pectoralis muscles that blocks the pectoral nerve as well as the long thoracic, intercostobrachial and lateral cutaneous branches of the inter-costal III, IV, V, and VI nerves. PECS-II is a less invasive and easier to be performed alternative to thoracic paravertebral block (TPVB). This block, defined by Blanco et al., provides safe and adequate post-operative analgesia in the anterior chest wall after breast surgery. The most common complications are pneumothorax, vascular puncture, infection, local anesthetic systemic toxicity (LAST), allergy and failed block .

ESPB is a paraspinal fascial plane block in which local anesthetic is injected between the tip of the transverse process of the spine and the anterior fascia of the erector spinae muscles blocking the dorsal and ventral rami of the spinal nerves, as well as the sympathetic chain, resulting in analgesia of chronic thoracic neuropathic pain, breast and upper abdominal surgeries. The block, defined by Forero et al., can cover several spinal nerve levels above and below the injection site as the local anesthetic spreads along the fascial plane, depending on the volume and concentration of the local anesthetic . The main advantages of this technique include the ease of performing it, the analgesic efficacy and the low risk of complications as Pneumothorax, hemi-diaphragmatic paralysis, motor weakness, and neurological findings related to local anesthesia toxicity .

ELIGIBILITY:
Inclusion Criteria:

1. Female patients scheduled for MRM.
2. Age eligible ≥ 40 & ≤ 65 yrs.
3. Patients with American Society of Anesthesiologists (ASA) physical status I, II who will be scheduled for Modified Radical Mastectomy surgery.

Exclusion Criteria:

1. Age < 40 & > 65 years old.
2. Declining to give written informed consent.
3. History of allergy to the medications used in the study.
4. Contraindication to regional anesthesia [including coagulopathy (platelet count ≤ 80,000, INR ≥ 1.5) and local infection].
5. Severe hepatic impairment (INR ≥ 1.5, Bilirubin ≥ 2, Albumin ≤ 2).
6. Renal dysfunction [GFR < 50 ml/min calculated by MDRD (Modification of diet in renal disease) equation for GFR estimation (Livio et al., 2008)].
7. Psychiatric disorder.
8. Pregnancy.
9. Patient with history of thoracic spine surgery.

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 20 (Actual)
Dates: Start 2024-06-01 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2024-12-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Ibrahim, MD, Principal Investigator — Faculty Of Medicine , Ain Shams University
Locations (1):
- Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Twenty patients were enrolled and randomly divided into the two groups , 10 patients each .
Groups:
- Modified Pectoral Plane Block Group: first group 10 patients
  Modified Pectoral Plane block group: The patient will lay supine with the ipsilateral arm abducted and externally rotated and the elbow flexed at 90 degrees. The probe will be placed transversely between the clavicle medially and above and the shoulder joint laterally. After identifying the pectoralis major and minor muscles and the plane between them, the probe will be pushed 1-2 cm caudally and medially. In a caudal tilt, within a biconvex space, the artery will be recognised. After that, the block needle will be inserted in an in-plane approach to the artery's location and 10 mL of 0.25% bupivacaine will be administered Then probe will be moved laterally and caudally towards the anterior axillary fold until the serratus muscle appears beneath the pectoralis minor muscle attaching to the underlying ribs. The needle will target the plane between pectoralis minor and serratus muscles at the level of the third rib, followed by negative aspiration into the fascial plane then injection of 10 mL of 0.25 bupivacaine.
Period: Overall Study
Arm/Group | Modified Pectoral Plane Block Group | Erector Spinae Plane Block Group
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Pectoral Plane Block Group: first group 10 patients
  Modified Pectoral Plane block group: The patient will lay supine with the ipsilateral arm abducted and externally rotated and the elbow flexed at 90 degrees. The probe will be placed transversely between the clavicle medially and above and the shoulder joint laterally. After identifying the pectoralis major and minor muscles and the plane between them, the probe will be pushed 1-2 cm caudally and medially. In a caudal tilt, within a biconvex space, the artery will be recognised. After that, the block needle will be inserted in an in-plane approach to the artery's location and 10 mL of 0.25% bupivacaine will be administered Then probe will be moved laterally and caudally towards the anterior axillary fold until the serratus muscle appears beneath the pectoralis minor muscle attaching to the underlying ribs. The needle will target the plane between pectoralis minor and serratus muscles at the level of the third rib, followed by negative aspiration into the fascial plane then injection of 10 mL of 0.25 bupivacaine.
- Total: Total of all reporting groups
Arm/Group | Pectoral Plane Block Group | Erector Spinae Plane Block Group | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.7 (1.9) | 52.1 (7.3) | 53.4 (5.33)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 10 | 20
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
weight [Mean (Standard Deviation); unit: kilograms] | 77.5 (7.8) | 72.8 (7) | 75.15 (7.41)
height [Mean (Standard Deviation); unit: centimeters] | 169.7 (3.9) | 167.8 (3.6) | 168.75 (3.75)
breast-side [Count of Participants; unit: Participants]
  unilateral | 8 | 7 | 15
  bilateral | 2 | 3 | 5
BMI [Mean (Standard Deviation); unit: kilogram per meter squared] | 26.9 (2.9) | 25.9 (3.0) | 26.4 (2.95)
ASA Classification [Number; unit: participants] — The American Society of Anesthesiologists (ASA) physical status classification system is a grading system to determine the health of a person before a surgical procedure that requires anesthesia where ASA I is a normal healthy patient ASA II a patient with mild systemic disease ASA III a patient with severe systemic disease ASA IV a patient with severe systemic disease that is a constant threat to life ASA V a moribund patient who is not expected to survive without the operation ASA VI a declared brain-dead patient whose organs are being removed for donor purposes
  participants
    ASA I = A normal healthy patient | 4 | 3 | 7
    ASA II = A patient with mild systemic disease | 6 | 7 | 13
operation duration [Mean (Standard Deviation); unit: minutes] | 113.4 (33.2) | 134.4 (15.8) | 123.9 (26)

OUTCOME MEASURES:

1. Primary Outcome: Post-operative Pain Severity Assessed by Visual Analogue Scale Immediately Postoperative on Admission to the Post Anesthesia Care Unit.
Description: Visual Analogue Scale is a scale for pain assessment ranging from 0 to 10 where 0 is minimum and means no pain while 10 is maximum and means maximum pain which means worse outcome
Time Frame: will be evaluated postoperatively on arrival to PACU (zero time)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Modified Pectoral Plane Block Group | Erector Spinae Plane Block Group
Number analyzed (Participants) | 10 | 10
score on a scale | 0.4 (0.5) | 0.9 (0.3)

2. Secondary Outcome: Post-operative Pain Severity Assessed by Visual Analogue Scale at 2 Hours, 4 Hours, 8 Hours, 12 Hours, 18 Hours and 24 Hours Post-operatively.
Description: Post-operative pain severity assessed by Visual analogue scale at 2 hours, 4 hours, 8 hours, 12 hours, 18 hours and 24 hours post-operatively where visual analogue scale ranges from zero to ten where (0 = no pain, 10 = maximum pain imaginable).
Time Frame: 24 hours post-operative
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pectoral Plane Block Group | Erector Spinae Plane Block Group
Number analyzed (Participants) | 10 | 10
score on a scale
  Post-operative pain severity assessed by Visual analogue scale at 2 hours postoperatively. | 1.3 (0.5) | 1.9 (0.3)
  Post-operative pain severity assessed by Visual analogue scale at 4 hours postoperatvely. | 1.4 (0.5) | 3.1 (0.3)
  Post-operative pain severity assessed by Visual analogue scale at 8 hours postoperatively. | 2.8 (0.6) | 3.8 (0.9)
  Post-operative pain severity assessed by Visual analogue scale at 12 hours postoperatively. | 2.5 (0.7) | 3.4 (1.1)
  Post-operative pain severity assessed by Visual analogue scale at 18 hours postoperatively. | 1.9 (0.6) | 2.9 (0.6)
  Post-operative pain severity assessed by Visual analogue scale at 24 hours postoperatively. | 1.6 (0.5) | 2 (0.5)

ADVERSE EVENTS:
Time Frame: 24 hours postoperative
Arm/Group | Modified Pectoral Plane Block Group | Erector Spinae Plane Block Group
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-08-01): https://cdn.clinicaltrials.gov/large-docs/82/NCT06714682/Prot_SAP_000.pdf